CLINICAL TRIAL: NCT04705935
Title: Amniochorionic Membrane Cells in the Maternal Blood as a Biomarker for Preterm Birth
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Arcedi Biotech (Industry); Aarhus University Hospital (Other); The University of Texas Medical Branch, Galveston (Other); Medical University of Graz (Other)
Responsible Party: Principal Investigator, Niels Uldbjerg, Professor, University of Aarhus
Other Study IDs: AU011020
Record Dates: First submitted 2020-12-01; First posted 2021-01-12 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Preterm Birth; Preterm Premature Rupture of Membrane; Preterm Labor
Keywords: Amniochorionic Membrane Cells; Fetal Membrane Cells
MeSH Terms: conditions — Premature Birth; Preterm Premature Rupture of the Membranes; Obstetric Labor, Premature

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (8):
- Term pregnant women without labor contractions or rupture of membranes: Term pregnant women > 37 weeks gestation with a normal pregnancy. One blood sample before a scheduled caesarean section.
- Term pregnant women with labor contractions: Term pregnant women > 37 weeks gestation with a normal pregnancy. One blood sample when labor contractions, but before spontaneous rupture of membranes.
- Term pregnant women with spontaneous rupture of membranes: Term pregnant women > 37 weeks gestation with a normal pregnancy. One blood sample after spontaneous rupture of membranes, but without labor contractions.
- Preterm labor contractions (PLC): One blood sample when labor contractions before 34 weeks gestation without rupture of membranes.
- Preterm Prelabor Rupture of the Fetal Membranes (PPROM): One blood sample when rupture of the fetal membranes before 34 weeks gestation without labor contractions.
- Control group: Women with normal pregnancies. One blood sample in gestation week 25+0 to 37 matched as controls for PLC and PPROM cases.
- Longitudinal cohort during pregnancy: Women with normal pregnancies, where blood samples will be collected at week 12, 20, 28, 34 and 36, as well as at labor.
- Longitudinal cohort post partum: Women with normal pregnancies, where blood samples will be collected at labor, as well as 2 days, and 4, 8 and 12 weeks after birth.

SUMMARY:
Globally, preterm birth (15 mill. per year) is the leading cause of under-5 child mortality (1 mill. per year) and morbidity. Important pathways include preterm labor contractions, Preterm Prelabor Rupture of the Fetal Membranes (PPROM), and iatrogenic delivery. At labor, the fetal amniochorionic membrane undergoes a cellular senescence and shed fetal amniochorionic membrane cells (ACM cells) to the maternal circulation. In collaboration with the private firm ARCEDI Biotech and The University of Texas Medical Branch at Galveston, Aarhus University has identified specific antibodies, which can be used to isolate ACM cells from maternal blood. Thus, the aim of this study is 1) to characterize ACM cells by histological and immunological techniques, and 2) in a cohort assess their performance as biomarkers of amniochorionic membrane dysfunction, including early detection of threatening preterm birth. In perspective, the findings are expected to improve the diagnostics and treatment of preterm birth.

DETAILED DESCRIPTION:
Aim:

The aim of the study is 1) to characterize circulating fetal amniochorionic membrane cells (ACM cells) in pregnant women and 2) to investigate if they can function as biomarkers of amniochorionic membrane dysfunction, including risk of preterm birth.

Background:

Globally, preterm birth (15 mill. per year) is the leading cause of under-5 child mortality (1 mill. per year) and morbidity. Important pathways include preterm labor contractions (PLC), Preterm Prelabor Rupture of the Fetal Membranes (PPROM), and iatrogenic delivery due to preeclampsia and fetal growth restriction.

At labor, the fetal amniochorionic membrane undergoes a cellular senescence and shed fetal amniochorionic membrane cells (ACM cells) to the maternal circulation. Similar features are expected to be seen in cases with PPROM. In collaboration with ARCEDI Biotech Aps and the University of Texas Medical Branch at Galveston, Aarhus University has identified specific fetal membrane cell markers, i.e. specific proteins highly expressed by the ACM cells. Commercially available antibodies specific for these identified proteins can be used to isolate ACM cells from the maternal blood. The preliminary studies indicate that circulating ACM cells are present in the second half of pregnancy but not in the first half of pregnancy.

The investigators want to confirm by immunohistochemistry that specific antibodies can identify ACM cells in the fetal membranes, and that they can be a platform for isolating ACM cells from the maternal circulation.

Materials and Methods:

The investigators will isolate ACM cells from maternal blood by Magnetic Activating Cell Sorting (MACS) using different specific antibodies for ACM cells. The enriched ACM cells will be stained using fluorescent-labeled cytokeratin and vimentin antibodies, and sorted individually by Fluorescence Activated Cell Sorting (FACS). The true identification of the fetal derived ACM cells will be done by Short Tandem Repeat (SRT) analysis.

The antibodies that perform best will be selected based on pilot studies on pregnant women at term and in gestation week 12, 20, 28 and 34, as well as at labor and post partum. The protein expression and specificity of each antibody will be confirmed by immunohistochemistry and bright field microscopy on biopsies from the fetal membranes, placental tissue, and the placental bed in the uterus.

The established protocol will be used to evaluate the number of ACM cells in the maternal blood in normal and pathological pregnancies on cross sectional cohorts of term pregnant women with and without labor contractions and spontaneous rupture of membranes, women with PLC before 34 weeks gestation, women with PPROM before 34 weeks gestation, and a control group at gestational age 25+0 to 37.

Perspectives:

In the future, the results are expected to improve the diagnostics and treatment of threatening preterm birth, thus preventing mortality and morbidity in millions of children worldwide.

ELIGIBILITY:
Inclusion Criteria:

* Normal pregnancy at term (> 37 weeks) the day before a planned caesarean section.
* Normal pregnancy at term (> 37 weeks) with planned vaginal delivery.
* Women with preterm labor contractions < 34 weeks admitted at the hospital.
* Women with PPROM < 34 weeks admitted at the hospital.
* Normal pregnancy at gestational age 25+0 to 37.
* Normal pregnancy at gestational age 12 included at the nuchal translucency scan.
* Normal pregnancy at birth.

Exclusion Criteria:

* Maternal age < 18
* Women who does not understand the oral or written information
* Women who does not speak Danish
* Women who does not want to participate
* Women with complications in pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Pregnant women who complies to the above mentioned inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2024-06-28 (Actual); Study Completion 2024-06-28 (Actual)

PRIMARY OUTCOMES:
ACM cells in maternal blood | At inclusion
  Number

SECONDARY OUTCOMES:
Gestational age at delivery | At delivery
  Weeks+days
Birth weight of child | At delivery
  Kg
APGAR score | At delivery
  <4, 4-7, or >7
Sex of child | At delivery
  M/F

OTHER OUTCOMES:
Maternal age | At inclusion
  Years
Maternal BMI | At inclusion
  kg/m

CONTACTS AND LOCATIONS:
Overall Officials: Ramkumar Menon, PhD, Study Chair — The University of Texas Medical Branch, Galveston; Torben Steiniche, DMSc, Study Chair — Aarhus University Hospital; Palle Schelde, MSc, Principal Investigator — Arcedi Biotech; Ripudaman Singh, PhD, Study Chair — Arcedi Biotech; Berthold Huppertz, PhD, Study Chair — Medical University of Graz
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-01): https://cdn.clinicaltrials.gov/large-docs/35/NCT04705935/Prot_SAP_000.pdf